CLINICAL TRIAL: NCT01342081
Title: A Double-masked Study of DE-111 Ophthalmic Solution Versus Tafluprost Ophthalmic Solution 0.0015% Alone and Concomitant Use of Tafluprost Ophthalmic Solution 0.0015% Plus Timolol Ophthalmic Solution 0.5% in Patients With Primary Open Angle Glaucoma or Ocular Hypertension -Phase 3, Confirmatory Study-
Brief Title: DE-111 Against Tafluprost Ophthalmic Solution 0.0015% Alone and Concomitant Use of Tafluprost Ophthalmic Solution 0.0015% Plus Timolol Ophthalmic Solution 0.5%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01111004
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary open angle glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): DE-111 ophthalmic solution
  Interventions: Drug: DE-111 ophthalmic solution
- 2 (Active Comparator): Tafluprost ophthalmic solution 0.0015%
  Interventions: Drug: Tafluprost ophthalmic solution 0.0015%
- 3 (Active Comparator): Concomitant use of tafluprost ophthalmic solution 0.0015% plus timolol ophthalmic solution 0.5%
  Interventions: Drug: Concomitant use of tafluprost ophthalmic solution 0.0015% plus timolol ophthalmic solution 0.5%

INTERVENTIONS:
Drug: DE-111 ophthalmic solution
  Arms: 1
Drug: Tafluprost ophthalmic solution 0.0015%
  Arms: 2
Drug: Concomitant use of tafluprost ophthalmic solution 0.0015% plus timolol ophthalmic solution 0.5%
  Arms: 3

SUMMARY:
DE-111 ophthalmic solution will be evaluated for superiority in comparison with Tafluprost 0.0015% ophthalmic solution, or for non-inferiority in comparison with Tafluprost 0.0015% and Timolol ophthalmic solution 0.5% used concomitantly, in IOP(intraocular pressure) -lowering effect in primary open-angle glaucoma or ocular hypertension patients, in a multicenter, randomized, double-masked, parallel-group comparison study. Safety will be compared and evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open angle glaucoma or ocular hypertension
* Provided signed, written informed consent
* 20 years of age and older
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Switched to following three arms randomly from Tafluprost ophthalmic solution 0.0015% (one drop at a time, once daily).
Groups:
- DE-111: DE-111 ophthalmic solution (one drop at a time, once daily) and Placebo ophthalmic solution (one drop at a time, BID) in both eyes.
- Tafluprost: Tafluprost ophthalmic solution 0.0015% (one drop at a time, once daily) and Placebo ophthalmic solution (one drop at a time, BID) in both eyes.
- Tafluprost Plus Timolol: Tafluprost ophthalmic solution 0.0015% (one drop at a time, once daily) and Timolol ophthalmic solution 0.5% (one drop at a time, BID) in both eyes.
Period: Overall Study
Arm/Group | DE-111 | Tafluprost | Tafluprost Plus Timolol
Started | 161 | 164 | 164
Completed | 159 | 162 | 163
Not Completed | 2 | 2 | 1
Not completed — Did not receive allocated intervention | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who have instilled the investigational drug at least once. Excluded from analysis in Tafluprost (n=1).
  Reason: Protocol Violation
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-111 | Tafluprost | Tafluprost Plus Timolol | Total
Number analyzed (Participants) | 161 | 163 | 163 | 487
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 92 | 81 | 87 | 260
  >=65 years | 69 | 82 | 76 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.6) | 63.0 (12.6) | 60.6 (13.6) | 61.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 95 | 81 | 252
  Male | 85 | 68 | 82 | 235
Region of Enrollment [Number; unit: participants]
  Japan | 161 | 163 | 163 | 487

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal IOP(Intraocular Pressure) at End of Study
Description: Mean diurnal IOP(intraocular pressure) was calculated as an average of IOP(intraocular pressure) at 9:30 (pre-dose), 11:30 and 17:30.
Time Frame: Week 0(Baseline) and Week 4(End of Study)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-111 | Tafluprost | Tafluprost Plus Timolol
Number analyzed (Participants) | 161 | 163 | 163
mmHg | -2.6 (1.8) | -0.9 (1.7) | -2.2 (1.8)
Statistical Analysis 1: Comparison: DE-111 vs Tafluprost; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.1 to -1.3]
Statistical Analysis 2: Comparison: DE-111 vs Tafluprost Plus Timolol; Non-inferiority was evaluated after superiority to tafluprost was confirmed; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 1.5 mmHg was used. Non-inferiority was claimed if the upper limit of the confidence interval of the difference is 1.5 mmHg or less; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.1]

ADVERSE EVENTS:
Time Frame: Week 0(Baseline) and Week 4(End of Study)
Description: 164 patients were allocated in Tafluprost + Timolol group, but, one patient of this group discontinued without dosing the investigational drug or control drug even once.
Arm/Group | DE-111 | Tafluprost | Tafluprost Plus Timolol
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/164 | 0/163
Other Adverse Events (participants affected / at risk) | 0/161 | 0/164 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No